CLINICAL TRIAL: NCT03656861
Title: Lithuanian Athletes' Aortic Root Diameter
Brief Title: Lithuanian Atletes' Aortic Diameter
Status: Completed | Type: Observational
Sponsor: Agne Slapsinskaite (Other)
Collaborators: Renata Žumbakytė-Šermukšnienė (Unknown); Baranauskaitė Miglė (Unknown); Berškienė Kristina (Unknown)
Responsible Party: Sponsor-Investigator, Agne Slapsinskaite, Principal Investigator, Institut Nacional d'Educacio Fisica de Catalunya
Organization: Institut Nacional d'Educacio Fisica de Catalunya (Other)
Other Study IDs: Kaunas Sport Medicine Centre
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Sports Accident; Athletes Heart
Keywords: Aortic Valve; Sinus of Valsalva; Echocardiography; Sudden cardiac death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes: 122 were athletes (41 females and 81 males). Of the 41 female athletes, 32 were endurance athletes, and 9 strength athletes. From 81 male athletes, 56 were endurance athletes, and 25 were strength athletes.
  Interventions: Other: Physical load
- Non-athletes: 29 were non-athletes (14 females and 15 males)

INTERVENTIONS:
Other: Physical load — The impact of training on cardiac structure and function depends on the type, intensity and duration of the activity, as well as previous physical activity engagement, genetics and gender type. More knowledge about cardiac pathophysiologic training adaptation is needed.
  Groups: Athletes

SUMMARY:
Recent developments in football have seen the sudden death of young football player due to aortic rupture hence reinforcing the controversy of football as a field with substantial risk for sudden cardiac arrest and death. Moreover, there is an argument that aortic dilatation and the subsequent event of thoracic aortic aneurysm may be an occupational disease due to the nature of some vocations (i.e., military and security personnel, blue collar workers, weightlifters, athletes etc.). Of particular importance, there is some evidence that elite athletic training is associated with small but significantly larger aortic root diameter. The purpose of this study was to investigate aortic root adaptation to physical workload and to determine if aortic root's and left ventricle sizes are contingent upon the physical workload

DETAILED DESCRIPTION:
A preliminary data was collected from a total of 944 subjects in Kaunas Sports Medicine Centre during the recruiting period in 2014-2015. Final data analysis consisted of 151 Caucasian subjects who met the inclusion criteria.

All subjects underwent two-dimensional (2D) transthoracic echocardiography (TTE) procedure. Prior to performing 2D TTE, subjects' arterial blood pressure, heart rate, height, weight, and self-reported physical activity levels were measured.

The Ultrasound system CX50 (Philips Ultrasound, Philips Healthcare, Philips Medical Systems Nederland, USA) - with transducer S5-1 was used in this study. Two physicians performed 2D TTE and averages for all variables of interest were computed. The measurements of aortic root and the left ventricle were drawn upon the guidelines of the American Society of Echocardiography and the European Association of Cardiovascular Imaging.

The maximal diameter of the sinuses of Valsalva was measured at end-diastole, in a strictly perpendicular plane to that of the long axis of the aorta using the edge to leading edge (L-L) convention. The aortic annulus was measured at midsystole from inner edge to inner edge (I-I). This was done in order to obtain the rounder shape and bigger diameter of aortic annulus.

ELIGIBILITY:
Inclusion Criteria:

* A total of 2D transthoracic echocardiography performed in Kaunas Sports Medicine Centre 2014-2015.
* Age range 16- 35 years, given the literature definition of 'young' and 'old' athletes as < 35 and > 35 years.
* Physical activity levels (athletes or non-athletes). Individuals who participated in sports for more than 4 years and 4.5 hours per week were included in the group of athletes. Individual who were active for less than 4 years and/or 4.5 hours per week were classified as non-athletes.
* Physical activity type (endurance and strength sports).
* No current or previous history cardiovascular diseases.
* No activity on the test day.
* Consent to participate in the study.

Exclusion Criteria:

* No 2D transthoracic echocardiography.
* Age below 16 or over 35.
* Involvement in sports for less than 4 years and 4.5 hours per week.
* Sports branches not included in the list of endurance or strength sports (i.e., sprint, high jump, etc.).
* Cardiovascular disease (i.e., hypertonic disease, Marfan syndrome, bicuspid aortic valve, detected cardiomyopathy, etc.).
* Physical activity on the echocardiography test day.
* No content to participate in the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The subjects were divided into groups according to gender (i.e., female, male), physical activity (i.e., athletes, non-athletes) and physical activity type (i.e., strength and endurance sports). Of the 151 subjects, 122 were athletes (41 females and 81 males) and 29 were non-athletes (14 females and 15 males). Of the 41 female athletes, 32 were endurance athletes, and 9 strength athletes. From 81 male athletes, 56 were endurance athletes, and 25 were strength athletes.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Measurement of aortic root at aortic valve annulus (AA) | Long-term adaptation more when 4 years of physical activity with 4.5 hours per week training sessions
  Changes in aortic root at aortic valve annulus (AA) and at individuals.
Measurement of aortic root at sinus of Valsalva (VS) | Long-term adaptation more when 4 years of physical activity with 4.5 hours per week training sessions
  Changes in aortic root at sinus of Valsalva (VS) individuals.

SECONDARY OUTCOMES:
Measurement of values of the left ventricle (LV): LV end-diastolic diameter (LVEDD) | Long-term adaptation more when 4 years of physical activity with 4.5 hours per week training sessions
  Changes values of the left ventricle (LV): LV end-diastolic diameter (LVEDD)
Measurement of values of interventricular septum thickness in diastole (IVSTd) | Long-term adaptation more when 4 years of physical activity with 4.5 hours per week training sessions
  Changes values of interventricular septum thickness in diastole (IVSTd)
LV posterior wall thickness in diastole (LVPWTd) | Long-term adaptation more when 4 years of physical activity with 4.5 hours per week training sessions
  Changes values of LV posterior wall thickness in diastole (LVPWTd)

IPD SHARING:
Plan to Share IPD: Undecided